CLINICAL TRIAL: NCT00647400
Title: A Multicenter Open-Label Continuation Study of the Long-term Safety and Efficacy of Adalimumab (D2E7) in Japanese Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Adalimumab in Adult Japanese Subjects With Psoriasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Abbott Japan Co.,Ltd (Industry); Eisai Co., Ltd. (Industry)
Responsible Party: Eiichi Makino, Abbott
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M04-702
Record Dates: First submitted 2008-03-27; First posted 2008-03-31 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

ARMS (2):
- Adalimumab 40 mg every other week (Experimental)
  Interventions: Biological: adalimumab
- Adalimumab 80 mg every other week (Experimental)
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — Adalimumab 40 mg every other week, subcutaneous
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab 40 mg every other week
Biological: adalimumab — Adalimumab 80 mg every other week, subcutaneous
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab 80 mg every other week

SUMMARY:
To evaluate efficacy, safety, and pharmacokinetics of adalimumab in Japanese participants with psoriasis

DETAILED DESCRIPTION:
This was a continuation trial of adalimumab in participants with moderate to severe chronic plaque psoriasis who had completed Study M04-688 (NCT00338754), a 24-week, double-blind, placebo-controlled study. This study was an open-label extension study that continued until the approval of adalimumab for the treatment of psoriasis in Japan.

During Study M04-688 (NCT00338754), participants received 24 weeks of treatment with adalimumab 40 mg every other week (eow) with or without a loading dose, adalimumab 80 mg eow, or placebo.

At the start of this study, participants who had received adalimumab 40 mg eow or adalimumab 80 mg eow in Study M04-688 (NCT00338754) continued on the same treatment regimen. Participants who had received placebo during Study M04-688 (NCT00338754) were re-randomized at the start of this study to receive adalimumab 40 mg eow or adalimumab 80 mg eow.

Participants in the adalimumab 40 mg eow treatment group who failed to achieve a PASI50 response (>= 50% reduction in the Psoriasis Area and Severity Index score from Baseline of Study M04-688 [NCT00338754]) at or anytime after Week 12 of this study were given the option to increase their dose to adalimumab 80 mg eow. Once the dose was escalated, there was no option to de-escalate dosing back to 40 mg eow. Participants who failed to achieve PASI50 responses while receiving adalimumab 80 mg eow may have been discontinued from the study after evaluating the risk/benefit of further treatment with adalimumab.

At Week 28 of this study, it was mandatory for all participants who started the study in the adalimumab 80 mg eow treatment group (i.e., not including the dose escalators described above) to reduce their dose to adalimumab 40 mg eow, regardless of their response status. Following this mandatory dose reduction, if these participants failed to achieve or maintain PASI50 response, they were permitted to escalate their dose to adalimumab 80 mg eow. There was no option to de-escalate dosing back to 40 mg eow following dose escalation.

Data in this clinical trial results disclosure are analyzed as observed according to treatment received at the start of this study (i.e., adalimumab 40 mg eow or adalimumab 80 mg eow) regardless of subsequent dose escalation. Data are summarized according to participants' cumulative exposure to adalimumab in Study M04-688 (NCT00338754) and this study.

ELIGIBILITY:
Inclusion Criteria:

- Participants who completed Study M04-688 (NCT00338754)

Exclusion Criteria:

- Participant is considered by the investigator, for any reason, to be an unsuitable candidate for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2006-04; Primary Completion 2007-09 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuko Kobayashi, Study Director — Abbott
Locations (64):
- Japan (64):
  - Site Ref # / Investigator 5491, Bunkyō City
  - Site Ref # / Investigator 5429, Chiyoda-ku
  - Site Ref # / Investigator 5464, Fukuoka
  - Site Ref # / Investigator 5477, Fukuoka
  - Site Ref # / Investigator 5492, Fukuoka
  - Site Ref # / Investigator 5504, Fukuoka
  - Site Ref # / Investigator 5400, Fukushima
  - Site Ref # / Investigator 5406, Fukushima
  - Site Ref # / Investigator 5407, Fukushima
  - Site Ref # / Investigator 5437, Fukushima
  - Site Ref # / Investigator 5401, Gifu
  - Site Ref # / Investigator 5434, Gifu
  - Site Ref # / Investigator 5408, Hamamatsu
  - Site Ref # / Investigator 5495, Hiroshima
  - Site Ref # / Investigator 5391, Hokkaido
  - Site Ref # / Investigator 5402, Ishikawa
  - Site Ref # / Investigator 5431, Itabashi-ku
  - Site Ref # / Investigator 5462, Kagoshima
  - Site Ref # / Investigator 5476, Kagoshima
  - Site Ref # / Investigator 5435, Kanagawa
  - Site Ref # / Investigator 5432, Kawachi-gun
  - Site Ref # / Investigator 5440, Kawasaki
  - Site Ref # / Investigator 5499, Kyoto
  - Site Ref # / Investigator 5503, Kyoto
  - Site Ref # / Investigator 5411, Minatoku
  - Site Ref # / Investigator 5404, Mitaka
  - Site Ref # / Investigator 5417, Miyagi
  - Site Ref # / Investigator 5463, Nagasaki
  - Site Ref # / Investigator 5427, Nagoya
  - Site Ref # / Investigator 5465, Nankoku
  - Site Ref # / Investigator 5493, Nankoku
  - Site Ref # / Investigator 5482, Nishinomiya
  - Site Ref # / Investigator 5395, Numakunai
  - Site Ref # / Investigator 5496, Okayama
  - Site Ref # / Investigator 5441, Osaka
  - Site Ref # / Investigator 5467, Osaka
  - Site Ref # / Investigator 5480, Osaka
  - Site Ref # / Investigator 5483, Osaka
  - Site Ref # / Investigator 5498, Osaka
  - Site Ref # / Investigator 5388, Sapporo
  - Site Ref # / Investigator 5396, Sapporo
  - Site Ref # / Investigator 5399, Sapporo
  - Site Ref # / Investigator 5414, Shinjuku-ku
  - Site Ref # / Investigator 5433, Shizuoka
  - Site Ref # / Investigator 5466, Suita
  - Site Ref # / Investigator 5497, Suita
  - Site Ref # / Investigator 5505, Suita
  - Site Ref # / Investigator 5481, Tokushima
  - Site Ref # / Investigator 5506, Tokushima
  - Site Ref # / Investigator 6918, Tokushima
  - Site Ref # / Investigator 5405, Tokyo
  - Site Ref # / Investigator 5409, Tokyo
  - Site Ref # / Investigator 5410, Tokyo
  - Site Ref # / Investigator 5412, Tokyo
  - Site Ref # / Investigator 5413, Tokyo
  - Site Ref # / Investigator 5430, Tokyo
  - Site Ref # / Investigator 6553, Tokyo
  - Site Ref # / Investigator 5468, Tsu
  - Site Ref # / Investigator 5475, Ube
  - Site Ref # / Investigator 5415, Urayasu
  - Site Ref # / Investigator 5438, Urayasu
  - Site Ref # / Investigator 5416, Yamagata
  - Site Ref # / Investigator 5403, Yokohama
  - Site Ref # / Investigator 5428, Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese participants with chronic plaque psoriasis who completed the blinded, placebo-controlled Study M04-688 (NCT00338754; 24-week duration) enrolled in the extension study, M04-702, an open-label study until adalimumab received approval for treatment of psoriasis in Japan.
Groups:
- Adalimumab 40 mg Every Other Week: Participants who had received adalimumab 40 mg eow during Study M04-688 (NCT00338754) or who had received placebo during Study M04-688 (NCT00338754) and were re-randomized to receive adalimumab 40 mg eow during this study.
- Adalimumab 80 mg Every Other Week: Participants who had received adalimumab 80 mg eow during Study M04-688 (NCT00338754) or who had received placebo during Study M04-688 (NCT00338754) and were re-randomized to receive adalimumab 80 mg eow during this study. All participants had to reduce their dosage to adalimumab 40 mg eow at Week 28 (after 52 or 28 weeks of total adalimumab exposure).
Period: Overall Study
Arm/Group | Adalimumab 40 mg Every Other Week | Adalimumab 80 mg Every Other Week
Started | 89 | 58
Completed | 67 | 45
Not Completed | 22 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab 40 mg Every Other Week | Adalimumab 80 mg Every Other Week | Total
Number analyzed (Participants) | 89 | 58 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 56 | 136
  >=65 years | 9 | 2 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 45.1 (13.39) | 42.9 (11.88) | 44.2 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 76 | 48 | 124
Region of Enrollment [Number; unit: participants]
  Japan | 89 | 58 | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 50% Reduction in PASI (Psoriasis Area and Severity Index) Score Compared With Baseline PASI Score (PASI50 Response)
Description: PASI scores range from 0 (best outcome) to 72 (worst outcome including erythema, induration, desquamation, and area affected). Baseline is defined as the last available PASI value prior to the first dose of study drug (adalimumab or placebo) in Study M04-688 (NCT00338754).
Time Frame: Baseline and 12, 24, 36, 52, 76, 100, 160, and 208 weeks after the first dose of adalimumab
Population: All participants enrolled in this study were included in this intent-to-treat (ITT) analysis. Results are presented as observed.
Measure: Number; unit: Participants
Arm/Group | Adalimumab 40 mg Every Other Week | Adalimumab 80 mg Every Other Week
Number analyzed (Participants) | 89 | 58
Participants
  12 weeks (N = 89 [40 mg eow] and 57 [80 mg eow]) | 78 | 54
  24 weeks (N = 88 [40 mg eow] and 56 [80 mg eow]) | 80 | 55
  36 weeks (N = 87 [40 mg eow] and 54 [80 mg eow]) | 79 | 52
  52 weeks (N = 85 [40 mg eow] and 52 [80 mg eow]) | 80 | 51
  76 weeks (N = 80 [40 mg eow] and 52 [80 mg eow]) | 76 | 52
  100 weeks (N = 78 [40 mg eow] and 52 [80 mg eow]) | 75 | 49
  160 weeks (N = 71 [40 mg eow] and 47 [80 mg eow]) | 71 | 47
  208 weeks (N = 29 [40 mg eow] and 14 [80 mg eow]) | 29 | 14

2. Secondary Outcome: Number of Participants With a 75% Reduction in PASI (Psoriasis Area and Severity Index) Score Compared With Baseline PASI Score (PASI75 Response)
Description: as for outcome 1
Time Frame: Baseline and 12, 24, 36, 52, 76, 100, 160, and 208 weeks after the first dose of adalimumab
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Adalimumab 40 mg Every Other Week | Adalimumab 80 mg Every Other Week
Number analyzed (Participants) | 89 | 58
Participants
  12 weeks (N = 89 [40 mg eow] and 57 [80 mg eow]) | 54 | 45
  24 weeks (N = 88 [40 mg eow] and 56 [80 mg eow]) | 69 | 50
  36 weeks (N = 87 [40 mg eow] and 54 [80 mg eow]) | 65 | 51
  52 weeks (N = 85 [40 mg eow] and 52 [80 mg eow]) | 67 | 48
  76 weeks (N = 80 [40 mg eow] and 52 [80 mg eow]) | 70 | 47
  100 weeks (N = 78 [40 mg eow] and 52 [80 mg eow]) | 66 | 43
  160 weeks (N = 71 [40 mg eow] and 47 [80 mg eow]) | 69 | 41
  208 weeks (N = 29 [40 mg eow] and 14 [80 mg eow]) | 27 | 13

3. Secondary Outcome: Number of Participants With a 90% Reduction in PASI (Psoriasis Area and Severity Index) Score Compared With Baseline PASI Score (PASI90 Response)
Description: as for outcome 1
Time Frame: Baseline and 12, 24, 36, 52, 76, 100, 160, and 208 weeks after the first dose of adalimumab
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Adalimumab 40 mg Every Other Week | Adalimumab 80 mg Every Other Week
Number analyzed (Participants) | 89 | 58
Participants
  12 weeks (N = 89 [40 mg eow] and 57 [80 mg eow]) | 31 | 29
  24 weeks (N = 88 [40 mg eow] and 56 [80 mg eow]) | 50 | 39
  36 weeks (N = 87 [40 mg eow] and 54 [80 mg eow]) | 54 | 44
  52 weeks (N = 85 [40 mg eow] and 52 [80 mg eow]) | 54 | 42
  76 weeks (N = 80 [40 mg eow] and 52 [80 mg eow]) | 55 | 38
  100 weeks (N = 78 [40 mg eow] and 52 [80 mg eow]) | 55 | 35
  160 weeks (N = 71 [40 mg eow] and 47 [80 mg eow]) | 57 | 33
  208 weeks (N = 29 [40 mg eow] and 14 [80 mg eow]) | 23 | 12

ADVERSE EVENTS:
Time Frame: Adverse events are reported starting from the first dose of adalimumab (in Study M04-688 [NCT00338754] or in Study M04-702) up to 70 days after the last dose of adalimumab.
Arm/Group | Adalimumab 40 mg Every Other Week | Adalimumab 80 mg Every Other Week
Serious Adverse Events (participants affected / at risk) | 19/89 | 11/58
Other Adverse Events (participants affected / at risk) | 88/89 | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg Every Other Week (N=89) | Adalimumab 80 mg Every Other Week (N=58)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Near drowning (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Miscarriage of partner (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg Every Other Week (N=89) | Adalimumab 80 mg Every Other Week (N=58)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 3
Palpitations (Cardiac disorders) | 1 | 3
Conjunctivitis (Eye disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 7
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4
Cheilitis (Gastrointestinal disorders) | 3 | 5
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 20 | 14
Gastritis (Gastrointestinal disorders) | 7 | 3
Gingival pain (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 6 | 5
Periodontitis (Gastrointestinal disorders) | 9 | 6
Stomach discomfort (Gastrointestinal disorders) | 1 | 4
Toothace (Gastrointestinal disorders) | 9 | 2
Vomiting (Gastrointestinal disorders) | 3 | 3
Adverse drug reaction (General disorders) | 7 | 10
Chest pain (General disorders) | 5 | 1
Feeling abnormal (General disorders) | 6 | 4
Injection site erythema (General disorders) | 16 | 4
Injection site pruritus (General disorders) | 4 | 3
Injection site reaction (General disorders) | 5 | 3
Injection site swelling (General disorders) | 2 | 3
Malaise (General disorders) | 12 | 8
Oedema peripheral (General disorders) | 7 | 4
Pain (General disorders) | 4 | 3
Pyrexia (General disorders) | 12 | 7
Swelling (General disorders) | 2 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 3
Hepatic steatotis (Hepatobiliary disorders) | 1 | 5
Seasonal allergy (Immune system disorders) | 6 | 5
Cystitis (Infections and infestations) | 3 | 3
Dental caries (Infections and infestations) | 18 | 6
Folliculitis (Infections and infestations) | 21 | 14
Furuncle (Infections and infestations) | 2 | 4
Herpes simplex (Infections and infestations) | 7 | 4
Hordeolum (Infections and infestations) | 4 | 3
Nasopharyngitis (Infections and infestations) | 67 | 45
Otitis media (Infections and infestations) | 2 | 5
Pharyngitis (Infections and infestations) | 6 | 7
Rhinitis (Infections and infestations) | 5 | 4
Tinea pedis (Infections and infestations) | 9 | 9
Upper respiratory tract infection (Infections and infestations) | 14 | 9
Arthropod sting (Injury, poisoning and procedural complications) | 10 | 2
Contusion (Injury, poisoning and procedural complications) | 9 | 3
Excoriation (Injury, poisoning and procedural complications) | 5 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 2
Alanine aminotransferase increased (Investigations) | 21 | 9
Antinuclear antibody increased (Investigations) | 21 | 8
Aspartate aminotransferase increased (Investigations) | 15 | 6
Bacteria urine identified (Investigations) | 8 | 2
Blood alkaline phosphatase increased (Investigations) | 6 | 1
Blood bilirubin increased (Investigations) | 9 | 4
Blood creatine phosphokinase increased (Investigations) | 21 | 15
Blood glucose increased (Investigations) | 5 | 6
Blood lactate dehydrogenase increased (Investigations) | 8 | 2
Blood triglycerides increased (Investigations) | 22 | 17
Blood uric acid increased (Investigations) | 13 | 11
Blood urine present (Investigations) | 12 | 5
C-reactive protein increased (Investigations) | 12 | 5
Eosinophil percentage increased (Investigations) | 6 | 2
Gamma-glutamyltransferase increased (Investigations) | 11 | 5
Glucose urine present (Investigations) | 7 | 3
Platelet count decreased (Investigations) | 5 | 0
Platelet count increased (Investigations) | 2 | 3
Protein urine present (Investigations) | 4 | 3
Weight decreased (Investigations) | 1 | 3
Weight increased (Investigations) | 6 | 5
White blood cell count increased (Investigations) | 7 | 2
White blood cells urine positive (Investigations) | 9 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 10 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 10
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 4
Shoulder pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Dizziness (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 19 | 8
Hypoaesthesia (Nervous system disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 10 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 | 8
Acne (Skin and subcutaneous tissue disorders) | 8 | 3
Asteatosis (Skin and subcutaneous tissue disorders) | 1 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 6 | 5
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1 | 6
Eczema (Skin and subcutaneous tissue disorders) | 10 | 10
Erythema (Skin and subcutaneous tissue disorders) | 6 | 9
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 3
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 9
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 6
Urticaria generalised (Skin and subcutaneous tissue disorders) | 0 | 3
Hypertension (Vascular disorders) | 6 | 5
Influenza (Infections and infestations) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements vary; the Medical Institution shall not disclose any material/information disclosed by Abbott Japan in connection with the Clinical Research or information obtained by conducting the Clinical Research to third parties without Abbott Japan's prior written approval. When Medical Institution intends to publish information obtained by conducting Clinical Research, Institution shall obtain Abbott Japan's prior written approval.